CLINICAL TRIAL: NCT06607497
Title: Better Risk Perception Via Patient Similarity to Control Hyperglycemia and Sustained by Telemonitoring
Acronym: BRILLIANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Collaborators: AISG Health Grand Challenge (Unknown)
Responsible Party: Principal Investigator, Tan Ngiap Chuan, Principal Investigator, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-2281
Record Dates: First submitted 2024-09-16; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): In arm 1, participants will attend the risk communication session utilizing AI module (PERDICT.AI) delivered by the study team integrated with Home-based Diabetes Monitoring (PTEC-DM) providing personalized guidance through teleconsultation in addition to usual care. Screen activity of PERDICT.AI will be recorded using a screen capture software. The entire session will be audio recorded.
  Interventions: Other: Intervention using an AI enabled risk communication tool (PERDICT.AI); Other: Telemonitoring with Primary Tech Enhanced Care (PTEC-DM)
- Arm 2 (Experimental): In arm 2, participants will attend the risk communication session utilising AI module (PERDICT.AI) without PTEC-DM. Screen activity of PERDICT.AI will be recorded using a screen capture software. The entire session will be audio recorded.
  Interventions: Other: Intervention using an AI enabled risk communication tool (PERDICT.AI)
- Arm 3 (No Intervention): Arm 3 will be the active control group, receiving only standard care

INTERVENTIONS:
Other: Intervention using an AI enabled risk communication tool (PERDICT.AI) — Risk communication using PERDICT.AI dynamically communicates an individual's glycemic control, offering a comparative ranking among peers to enhance motivation and awareness. Furthermore, it assesses the risk of potential complications comparing with peer data with exemplary cases to underscore the consequences of suboptimal management. In addition, it will generate personalized recommendations including medication adjustment and personalized health plans.
  Arms: Arm 1; Arm 2
Other: Telemonitoring with Primary Tech Enhanced Care (PTEC-DM) — The Primary Tech-Enhanced Care (PTEC) programme focuses on encouraging patients to manage chronic conditions at home through user-friendly kits. The Home Diabetes Monitoring programme (PTEC-DM) enables home-based glucose and blood pressure monitoring once a week using a Bluetooth enabled device. These reading will be securely transmitted to the study team via the app and managed appropriately through teleconsultation. Additionally, participants will receive health nudges, encouragements, and reminders through in-app messages to support their well-being.
  Arms: Arm 1

SUMMARY:
Background: Diabetes significantly raises the likelihood of complications, thereby increasing the risk of diabetes-related mortality, particularly due to vascular complications. It is vital to address this rising trend of mortality, by enhancing awareness of diabetes complications to improve risk perception and ultimately reduce mortality rates. Managing diabetes effectively requires interventions addressing both risk communication and monitoring, helping patients better understand and make informed decisions about their health.

Objectives: The primary aim is to evaluate and compare the effectiveness of combined risk communication session using an AI module (PERDICT.AI) and home-based diabetes monitoring (PTEC-DM) versus a standalone risk communication session in improving health outcomes (risk perception, medication adherence, self-care activities and glycaemic control) among poorly controlled diabetes patients. Secondary aims are to explore participants' views and experiences of risk communication session using PERDICT.AI, PTEC-DM and usual care and clinician' views on utility of the new approach to improve risk perception.

Methods: A mixed-method study design will be employed to conduct a multi-arm randomized controlled trial across four of the SingHealth Polyclinics cluster (Pasir Ris, Eunos, Sengkang, Tampines North). Patient participants will be randomly allocated in a 1:1:1 ratio to one of the three arms. Arm 1 will receive risk communication session using PERDICT.AI and home-based diabetes monitoring using PTEC-DM alongside usual care. Arm 2 participants will undergo a standalone risk communication session using PERDICT.AI with usual care while arm 3 will serve as the control group with usual care. A total of 360 (120 in each group) participants will be enrolled by simple randomization. Eligible patient must be of age between 36 and 65 years with HbA1c >8.0% within the last 6 months.

Significance of the study: Findings from the study may add evidence to the scientific knowledge of using these approaches to improve risk perception and recommend development of similar interventions.

DETAILED DESCRIPTION:
Diabetes has emerged as a significant public health concern globally, and Singapore is no exception. As of 2022, 8.5% of the adults in Singapore is affected by diabetes and the number is expected to reach 1 million by 2050, making it imperative to address the associated challenges. The economic implications of diabetes extend beyond healthcare costs, impacting productivity and quality of life. The total cost among the working-age population with diabetes - direct and indirect costs included - is expected to rise from USD 787 million (USD 5,646 per person) in 2010 to USD 1,867 million in 2050 (USD 7,791 per person).

In addition, diabetes poses a substantial risk of complications that can adversely impact various organ systems. Complications such as cardiovascular diseases, neuropathy, and retinopathy pose severe threats to the health of individuals with poorly managed diabetes. A study on global trend of diabetes mortality revealed a concerning global increase in diabetes-related mortality, particularly due to vascular complications, posing a significant challenge to diabetes management. To address the rising trends of mortality, it is crucial to enhance awareness of diabetes complications to improve risk perception and ultimately reduce mortality rates.

Perceived risk of diabetes complications can impact patient behavior, influencing adherence to treatment plans and lifestyle changes. Individuals with a higher risk perception may be more likely to engage in proactive management, leading to better health outcomes and potentially reducing mortality rates associated with diabetes complications. On the other hand, individuals with poorer risk perception may neglect necessary precautions, leading to suboptimal disease management and an increased likelihood of complications, potentially impacting mortality rates.

A systematic review on risk perceptions of diabetes complications highlights a concerning lack of awareness regarding the risk of diabetes related complications among individuals with type 2 diabetes mellitus (T2DM). Similarly, research studies on diabetes complications risk awareness, particularly in Singapore, revealed knowledge gaps among adults. Despite the significant impact on quality of life, later-stage T2DM and its complications were perceived as slowly progressing and not immediately life-threatening. Hence, for poorly controlled diabetes patients, effective communication regarding the risks of complications is paramount.

Weaver et al defined risk communication as "the effective and accurate exchange of information about health risks and hazards" so as to "advance risk awareness and understanding and promote health-protective behaviors". Enhancing risk communication not only promotes informed decision-making but also advances early intervention and preventive measures. Furthermore, Hashim J et al emphasized the importance of considering social and cultural factors in the development of effective interventions among adults with elevated risk perception yet do not engage in preventive actions. The study also suggested that diverse perspectives concerning the benefits and weaknesses related to preventive measures can impact the long-term sustainability of these behaviors.

Risk communication interventions have been developed for patients with T2DM to improve their risk perceptions and health actions. These interventional studies explore different methods to communicate diabetes complication risks to those with T2DM. interventions include range of innovative risk communication methods like visual aids, general nudges, digital tool for personalized risk information and family support through WeChat. While such interventions contribute to valuable insights, there are some limitations with these tools like limited long-term impact, technology adoption challenges. Addressing these drawbacks with an integrated approach could enhance the robustness and applicability of the findings in diverse healthcare settings.

PERDICT.AI based counselling

An AI-enabled similarity-based model, named PERDICT.AI (Personalised Diabetes Counselling Tool using Artificial Intelligence) was developed by a team of primary care physicians and computer scientists in Singapore to help physicians communicate risks to patients with diabetes mellitus. The tool ranks a patients' HbA1c levels with similar patients (or peers) from a de-identified database, showing how prevalent diabetes complications are based on HbA1c severity. This is referred to as "peer-comparison" and the tool underwent revisions following feedback from primary care physicians to enhance its usefulness in risk communication.

Based on Health Belief Model (HBM), a risk communication intervention, was developed for Primary care Physicians (PCPs) to counsel patients with T2DM on their glycemic control and the complications that could arise, and to recommend ways to improve glycemic control and prevent complications (or further complications). This will be supported by information from PERDICT.AI.

Risk communication using PERDICT.AI dynamically communicates an individual's glycaemic control, offering a comparative ranking among peers to enhance motivation and awareness. Furthermore, it assesses the risk of potential complications comparing with peer data with exemplary cases to underscore the consequences of suboptimal management. In addition, it will generate personalized recommendations including medication adjustment and personalized health plans.

Diabetes management often requires consistent encouragement and guidance, which a static risk communication tool may not deliver. In addition, passive receipt of information might not motivate patients to actively take part in diabetes management. Such lack of engagement could lead to reduced adherence to recommended strategies, limiting the tool's overall impact. This is evident from the @RISK study, where the improved risk perception observed initially at 2 weeks dissipated by the 12th week, highlighting a temporal limitation in sustaining positive outcomes. Although participants in the intervention arm reported higher satisfaction with risk communication, this did not translate into sustained improvements. This underscores the need for an integrated approach to sustain positive outcomes beyond short-term.

Integration with telemonitoring system

Sustaining improved risk perception over an extended period can be achieved through telemonitoring. By utilizing telemonitoring technology, healthcare providers can maintain a consistent connection with patients, offering real-time insights into their health status. Additionally, telemonitoring facilitates continuous education and support, thereby contributing to the long-term sustainability of improved risk perception and can significantly enhance diabetes management and prevent complications.

The Primary Tech-Enhanced Care (PTEC) programme focuses on encouraging patients to manage chronic conditions at home through user-friendly kits. The Home Diabetes Monitoring programme (PTEC-DM) enables home-based glucose and blood pressure monitoring once a week using a Bluetooth enabled device. These reading will be securely transmitted to the study team via the app and managed appropriately through teleconsultation. Additionally, participants will receive health nudges, encouragements, and reminders through in-app messages to support their well-being.

The integration of PTEC-DM with the risk communication using PERDICT.AI capitalizes on the strengths of human interaction and adaptability, contributing to a more holistic and patient-centred diabetes management approach. Such combined approach addresses both monitoring and guidance, contributing to enhanced patient understanding and informed decision-making. Hence this study is designed with the following objectives, adopting a multi-site, multi-arm randomized controlled trial design.

Objectives

Primary objective:

i. To assess the effectiveness of the risk communication using an AI enabled tool (PERDICT.AI) in improving risk perception score, quality of life and health outcomes (medication adherence and selfcare activities and glycemic control) among poorly controlled diabetes patients ii. To determine the effectiveness of a combination of risk communication session using PERDICT.AI and telemonitoring (PTEC-DM) in improving risk perception, quality of life and health outcomes

Secondary objectives:

iii. To compare the impact of the two approaches in improving risk perception, quality of life and health outcomes among poorly controlled diabetes patients iv. To assess the cost-effectiveness of the advanced care by comparing the incremental costs and health outcomes v. To explore participants' views and experiences of risk communication session using PERDICT.AI, PTEC-DM and usual care vi. To explore clinician' views on utility of the new approach to improve risk perception

Hypothesis:

• There will be improvement in patients' risk perception score and health outcomes (glycemic control and self-care activities) after the intervention.

Materials and methods

Study setting The study will be conducted at 4 polyclinics from a primary care clinic cluster taking care of more than 200,000 residents with diabetes in the Eastern region of Singapore.

Study design Sequential explanatory mixed-method study

Quantitative: Multi-arm randomized controlled trial (RCT) at four polyclinics which includes SingHealth Polyclinics at Pasir Ris, Tampines North, Eunos and Sengkang.

Qualitative: In-depth interview among the study participants' and clinician, who are integral part of the study team delivering interventions.

Quantitative: Multi-arm RCT This RCT involves three arms, incorporating a combination of interventions and standard care, as outlined below.

Arm 1: Advanced care with risk communication using an AI enabled tool (PERDICT.AI) + home-based monitoring using PTEC DM (main intervention arm) Arm 2: Usual care + risk communication using an AI enabled tool (PERDICT.AI) Arm 3: Usual care All groups will also receive a diabetes pamphlet.

Randomization Patient participants from each study site will be randomly allocated in a 1:1:1 ratio to one of the above-mentioned arms in an open-label fashion, using computer-generated random numbers for simple randomization of subjects. The nature of the intervention makes impossible to blind patients and research team to participant allocation. The randomization sequence is written and kept in an opaque sealed envelope, which will be labelled with a serial number. The study team will open the sealed envelope once the patient has consented to participate and then will be assigned to the study arms accordingly. All participants will receive a diabetes pamphlet ('Pamphlet - Taking Control of Diabetes').

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus on follow-up at the study site for at least 12 months
* Age 36 to 65 years
* At least one HbA1c reading ≥ 8.0% within the last 6 months
* Able to read and speak English

Exclusion Criteria:

* Not a Singapore citizen or permanent resident
* Pregnant
* End-stage kidney disease or on renal replacement therapy
* Known terminal illness
* Visual and/or hearing impairment
* Cognitive impairment or mental illness
* Unable to provide informed consent

Ages: 36 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Risk Perception Survey-Diabetes Mellitus (RPS-DM) | through study completion, an average of 12 to 16 months
  The RPS-DM consists of 31 questions. The first section assesses risk knowledge (5 items scored on 3-point scale with 1 point for each correct answer; higher score indicates greater knowledge of the risk of getting diabetes complications). The remaining 26 items comprise 5 subscales which can be described as: perceived personal control (4 items scored on 4-point scale); worry (2 items scored on 4-point scale), optimistic bias (2 items scored on 4-point scale); personal disease risk (9 items scored on a 4-point scale; indicates degree of own perceived risk of getting 9 diseases or conditions, plus additional question about whether they have ever had the condition, scored yes/no with 1 point added for yes response); and environmental risk (9 items scored on a 4-point scale). The composite risk perception is the average of the 26 items in the main questionnaire; higher scores indicate greater comparative perceived risk.
Health related Quality of life | through study completion, an average of 12 to 16 months
  Change in the scores using EQ-5D-5L questionnaire; The EQ-5D-5L tool comprises five dimensions, each describing a different aspect of health: mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression. Each dimension has five response levels (no problems, slight problems, moderate problems, severe problems, unable to/ extreme problems). The proportion of patients reporting each level of problem on each dimension of the EQ-5D will be determined through study completion and compared. EQ VAS (Visual Analogue Scale) provides a quantitative measure of the patient's perception of their overall health. The EQ VAS records the respondent's overall current health on a vertical scale (0-100), where the endpoints are labelled '0-The worst health you can imagine' and '100-The best health you can imagine'.
Medication adherence | through study completion, an average of 12 to 16 months
  Change in the scores using five item Medication Adherence Report Scale (MARS-5); MARS-5 score was calculated by summing the numeric score (range 1-5) from each question for out of 25 (range 5-25). A higher score indicates better adherence.
Summary of Diabetes Self-care Activities (SDSCA) questionnaire | through study completion, an average of 12 to 16 months
  SDSCA questionnaire collects data on general diet, specific diet, exercise, blood-glucose testing, foot care, and smoking, using an 8-point Likert-type scale (0-7), which represents the number of days per week when the given self-care activity was performed. Scores are calculated separately for each item and the level of adherence is indicated by the mean score for each dimension.
Iowa-Netherlands Comparison Orientation Measure (INCOM) | baseline enrolment
  The INCOM is an 11-item measure of one's tendency to make social comparisons. The scale includes such items as: "I always like to know what others in a similar situation would do." Response choices range from 1 (disagree strongly) to 5 (agree strongly). Higher scores indicate more of a tendency to socially compare.

SECONDARY OUTCOMES:
Cost-effectiveness analysis | through study completion, an average of 12 to 16 months
  Unit costs for consultation, laboratory, hospitalization, and pharmacy services, as well as the expenses for home-based monitoring (including a Bluetooth-enabled glucometer, test strips, lancets, and a blood pressure monitor), will be estimated to assess the cost-effectiveness of the advanced care by comparing the incremental costs and health outcomes
Views and experiences of risk communication session using PERDICT.AI, PTEC-DM and usual care | 24-48 weeks
  in-depth interview with the participants till point of data saturation
Exploring clinician' views on utility of combined intervention to improve risk perception | 24-48 weeks
  in-depth interview with the study team doctors till point of data saturation

CONTACTS AND LOCATIONS:
Overall Officials: Ngiap Chuan Tan, MMed, Principal Investigator — SingHealth Polyclinics
Locations (1):
- SingHealth Polyclinics, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Png ME, Yoong J, Phan TP, Wee HL. Current and future economic burden of diabetes among working-age adults in Asia: conservative estimates for Singapore from 2010-2050. BMC Public Health. 2016 Feb 16;16:153. doi: 10.1186/s12889-016-2827-1. PMID 26880337
- [Background] Ling W, Huang Y, Huang YM, Fan RR, Sui Y, Zhao HL. Global trend of diabetes mortality attributed to vascular complications, 2000-2016. Cardiovasc Diabetol. 2020 Oct 20;19(1):182. doi: 10.1186/s12933-020-01159-5. PMID 33081808
- [Background] Nie R, Han Y, Xu J, Huang Q, Mao J. Illness perception, risk perception and health promotion self-care behaviors among Chinese patient with type 2 diabetes: A cross-sectional survey. Appl Nurs Res. 2018 Feb;39:89-96. doi: 10.1016/j.apnr.2017.11.010. Epub 2017 Nov 7. PMID 29422183
- [Background] Mousavizadeh SN, Ashktorab T, Ahmadi F, Zandi M. From Negligence to Perception of Complexities in Adherence to Treatment Process in People with Diabetes: A Grounded Theory Study. Iran J Med Sci. 2018 Mar;43(2):150-157. PMID 29749983
- [Background] Rouyard T, Kent S, Baskerville R, Leal J, Gray A. Perceptions of risks for diabetes-related complications in Type 2 diabetes populations: a systematic review. Diabet Med. 2017 Apr;34(4):467-477. doi: 10.1111/dme.13285. Epub 2016 Nov 29. PMID 27864886
- [Background] Wee HL, Ho HK, Li SC. Public awareness of diabetes mellitus in Singapore. Singapore Med J. 2002 Mar;43(3):128-34. PMID 12005338
- [Background] Tham KY, Ong JJ, Tan DK, How KY. How much do diabetic patients know about diabetes mellitus and its complications? Ann Acad Med Singap. 2004 Jul;33(4):503-9. PMID 15329765
- [Background] Hashim J, Smith HE, Tai ES, Yi H. Lay perceptions of diabetes mellitus and prevention costs and benefits among adults undiagnosed with the condition in Singapore: a qualitative study. BMC Public Health. 2022 Aug 20;22(1):1582. doi: 10.1186/s12889-022-14020-z. PMID 35987615
- [Background] Welschen LM, Bot SD, Dekker JM, Timmermans DR, van der Weijden T, Nijpels G. The @RISK Study: Risk communication for patients with type 2 diabetes: design of a randomised controlled trial. BMC Public Health. 2010 Aug 5;10:457. doi: 10.1186/1471-2458-10-457. PMID 20687924
- [Background] Welschen LM, Bot SD, Kostense PJ, Dekker JM, Timmermans DR, van der Weijden T, Nijpels G. Effects of cardiovascular disease risk communication for patients with type 2 diabetes on risk perception in a randomized controlled trial: the @RISK study. Diabetes Care. 2012 Dec;35(12):2485-92. doi: 10.2337/dc11-2130. Epub 2012 Aug 24. PMID 22923669
- [Background] Rouyard T, Leal J, Baskerville R, Velardo C, Salvi D, Gray A. Nudging people with Type 2 diabetes towards better self-management through personalized risk communication: A pilot randomized controlled trial in primary care. Endocrinol Diabetes Metab. 2018 Jun 22;1(3):e00022. doi: 10.1002/edm2.22. eCollection 2018 Jul. PMID 30815556
- [Background] Rouyard T, Leal J, Salvi D, Baskerville R, Velardo C, Gray A. An Intuitive Risk Communication Tool to Enhance Patient-Provider Partnership in Diabetes Consultation. J Diabetes Sci Technol. 2022 Jul;16(4):988-994. doi: 10.1177/1932296821995800. Epub 2021 Mar 3. PMID 33655766
- [Background] Mao L, Lu J, Zhang Q, Zhao Y, Chen G, Sun M, Chang F, Li X. Family-based intervention for patients with type 2 diabetes via WeChat in China: protocol for a randomized controlled trial. BMC Public Health. 2019 Apr 5;19(1):381. doi: 10.1186/s12889-019-6702-8. PMID 30953483
- [Background] Feng Y, Zhao Y, Mao L, Gu M, Yuan H, Lu J, Zhang Q, Zhao Q, Li X. The Effectiveness of an eHealth Family-Based Intervention Program in Patients With Uncontrolled Type 2 Diabetes Mellitus (T2DM) in the Community Via WeChat: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2023 Mar 20;11:e40420. doi: 10.2196/40420. PMID 36939825
- [Background] Fang HSA, Tan NC, Tan WY, Oei RW, Lee ML, Hsu W. Patient similarity analytics for explainable clinical risk prediction. BMC Med Inform Decis Mak. 2021 Jul 1;21(1):207. doi: 10.1186/s12911-021-01566-y. PMID 34210320
- [Background] Oei RW, Fang HSA, Tan WY, Hsu W, Lee ML, Tan NC. Using Domain Knowledge and Data-Driven Insights for Patient Similarity Analytics. J Pers Med. 2021 Jul 22;11(8):699. doi: 10.3390/jpm11080699. PMID 34442343
- [Background] Andres E, Meyer L, Zulfiqar AA, Hajjam M, Talha S, Bahougne T, Erve S, Hajjam J, Doucet J, Jeandidier N, Hajjam El Hassani A. Telemonitoring in diabetes: evolution of concepts and technologies, with a focus on results of the more recent studies. J Med Life. 2019 Jul-Sep;12(3):203-214. doi: 10.25122/jml-2019-0006. PMID 31666818
- [Background] Lim DYZ, Chia SY, Abdul Kadir H, Mohamed Salim NN, Bee YM. Establishment of the SingHealth Diabetes Registry. Clin Epidemiol. 2021 Mar 16;13:215-223. doi: 10.2147/CLEP.S300663. eCollection 2021. PMID 33762850
- [Background] Gibbons FX, Buunk BP. Individual differences in social comparison: development of a scale of social comparison orientation. J Pers Soc Psychol. 1999 Jan;76(1):129-42. doi: 10.1037//0022-3514.76.1.129. PMID 9972558
- [Background] Walker EA, Caban A, Schechter CB, Basch CE, Blanco E, DeWitt T, Kalten MR, Mera MS, Mojica G. Measuring comparative risk perceptions in an urban minority population: the risk perception survey for diabetes. Diabetes Educ. 2007 Jan-Feb;33(1):103-10. doi: 10.1177/0145721706298198. PMID 17272796
- [Background] Seng JJB, Kwan YH, Fong W, Phang JK, Lui NL, Thumboo J, Leung YY. Validity and reliability of EQ-5D-5L among patients with axial spondyloarthritis in Singapore. Eur J Rheumatol. 2020 Apr;7(2):71-78. doi: 10.5152/eurjrheum.2020.19043. Epub 2020 Apr 1. PMID 32644927
- [Background] Chan AHY, Horne R, Hankins M, Chisari C. The Medication Adherence Report Scale: A measurement tool for eliciting patients' reports of nonadherence. Br J Clin Pharmacol. 2020 Jul;86(7):1281-1288. doi: 10.1111/bcp.14193. Epub 2020 May 18. PMID 31823381
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844